CLINICAL TRIAL: NCT04277143
Title: The Influence Factors of Pharmacokinetics/Pharmacodynamics of Daptomycin in Severe Patients and the the Effect of Different Blood Concentration of Daptomycin on the Outcomes of Renal Function
Brief Title: A Pharmacokinetics Study of Daptomycin in Critically Ill Patients and Effects of Daptomycin on Kidney
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, ZhiYong Peng, Professor; Chief physician, Zhongnan Hospital
Other Study IDs: 2019018
Record Dates: First submitted 2020-02-16; First posted 2020-02-20 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Outcome, Fatal; Infection
Keywords: daptomycin; pharmacokinetics; pharmacodynamics; critical ill patients; outcome
MeSH Terms: conditions — Infections | interventions — Daptomycin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Take blood and urine samples at several time points before and after daptomycin administration, and measure the blood and urine concentrations of the patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- critical ill patient with bloodstream infections: Severe patients with bloodstream infections often have sepsis / septic shock, acute kidney injury (AKI), hypoproteinemia, and renal replacement treatment.
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — Adult patients are given the recommended dose of daptomycin for injection. Patients with creatinine clearance (CLCR) ≥ 30 mL / min: 6 mg / kg every 24 hours.
  Patients with creatinine clearance (CLCR) <30mL / min (including hemodialysis or peritoneal dialysis): 6mg / kg every 48 hours. Dissolve 6mg / kg of this drug in 0.9% sodium chloride injection and instill it over a 30-minute time course once every 24 or 48 hours.

SUMMARY:
Daptomycin ，is the ﬁrst approved member of a new class of antimicrobials, the cyclic lipopeptides, and presents selective action against gram-positive bacteria, including methicillin- and vancomycin-resistant strains，disrupting the transfer of amino acids in the cell membrane, thus hindering the biosynthesis of bacterial cell cell wall peptide polysaccharide, changing the properties of cytoplasm membrane, can destroy bacterial cell membrane function in many ways, and quickly kill gram-positive bacteria. Because of its unique chemical structure and sterilization mechanism, bacteria rarely develop resistance to daptomycin. Daptomycin can be reversibility combined with human plasma protein (mainly serum albumin) and metabolized mainly through the kidneys.

There is still a lot of controversy about the application of daptomycin in patients with severe illness. Although studies suggest that daptomycin has less damage to kidney function than vancomycin, the effect of daptomycin on kidney function in severely ill patients is not yet clear, and more clinical studies are needed to explore their relationship. In addition, it is not clear whether the physiological pathology of specific populations such as sepsis/infectious shock, acute kidney injury, (AKI), hypoproteinemia, and renal replacement treatment affects the pharmacokinetics/pharmacodynamics of Daptomycin.

By exploring the application of daptomycin in patients with severe illness, this study explores the effects of special pathological physiological states such as sepsis/infectious shock and hypoproteinemia on daptomycin PK/PD, as well as the effects of different hemoglobin concentrations of daptomycin on the outcome of kidney function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severe bloodstream infections eligible for daptomycin indications
2. Treatment in the ICU
3. Patients aged 18 to 65

Exclusion Criteria:

1. Pregnant and lactating women
2. The patient or his agent refused to participate in the trial
3. Incomplete clinical medical information
4. Patient participates in another clinical trial at the same time
5. Previous history of myopathy or current CPK increase more than 2 times than normal
6. Patients need to use warfarin anticoagulation
7. Patients use tobramycin for anti-infection
8. Patients use drugs such as cyclosporine and fibrates that can cause adverse reactions to muscle disease
9. Patients with Gram-negative bacterial infections caused by abdominal and respiratory infections
10. Patients with heart failure, respiratory failure, Glasgow coma index (GCS) ≤ 8 points, liver function CHILD PUGH score C that are not related to the infection

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Department of Critical Medicine, Zhongnan Hospital of Wuhan University , considering bloodstream infections caused by Gram-positive bacteria。
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Apparent volume of distribution | 1 week
  Apparent volume of distribution of daptomycin in the patient's blood
Peak plasma concentration | 1 week
  Peak plasma concentration of daptomycin
Plasma trough concentration | 1 week
  Plasma trough concentration of daptomycin
Area under the plasma concentration versus time curve (AUC) | 1 week
  Area under the plasma concentration versus time curve (AUC) of daptomycin
Clearance of daptomycin | 1 week
  Daptomycin is metabolized mainly by the kidneys
Half-life | 1 week
  Half-life of plasma daptomycin
Protein binding rate | 1 week
  Reversible binding of daptomycin to plasma proteins (mainly serum albumin)
Serum creatinine | 1 week
  Serum creatinine can reflect kidney function
Urine output | 1 week
  Urine volume can reflect kidney function
Blood Urea Nitrogen | 1 week
  It can reflect kidney function
Urine protein | 1 week
  Reflect kidney function
Cystatin C | 1 week
  Reflect kidney function
β2-microglobulin(β2-MG) | 1 week
  Reflect kidney function
Major Adverse kidney Event（MAKE） | 28days
  Major Adverse kidney Event（MAKE）Refers to death, need for renal replacement therapy, and creatinine levels that are twice or more the baseline value；It can reflects the outcome of renal function.
ICU mortality | 28days
  Reflect patient prognosis
In-hospital mortality | 28days
  Reflect patient prognosis
ICU hospital stay length | 28 days
  Reflect patient prognosis
Total hospital stay length | 28 days
  Reflect patient prognosis

SECONDARY OUTCOMES:
White blood cell count | 1 week
  Reflect the severity of the patient's infection
Neutrophil ratio | 1 week
  Reflect the severity of the patient's infection
C-Reactive Protein | 1 week
  Reflect the severity of the patient's infection
Procalcitonin | 1 week
  Reflect the severity of the patient's infection
Interleukin-6 | 1 week
  Reflect the severity of the patient's infection
Bacterial culture results | 1 week
  Reflect the severity of the patient's infection
Body temperature | 1 week
  Reflect the severity of the patient's infection
Vascular drug use days | 1 week
  Assess patients' systemic circulation

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Peng, Professor, Principal Investigator — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No